CLINICAL TRIAL: NCT01286194
Title: A Multi-Center, Open-Label, All-Comers, Single Group Observational Study to Investigate Use Patterns and Safety in Simulated Actual Over-the-counter (OTC )Use of Rabeprazole Sodium for the Treatment of Heartburn Symptoms
Brief Title: A Study to Investigate Use Patterns and Safety in Simulated Actual Over-the-counter (OTC) Use of Rabeprazole Sodium for the Treatment of Heartburn Symptoms
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Marco Cyrille, MD, Eisai, Inc
Other Study IDs: E3810-A001-315
Record Dates: First submitted 2011-01-11; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2006-01

CONDITIONS: Frequent Heartburn
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Experimental 1
  Interventions: Drug: Rabeprazole sodium

INTERVENTIONS:
Drug: Rabeprazole sodium — Rabeprazole sodium 10 mg orally every day for 14 days

SUMMARY:
This is a multi-center, open-label, all-comers OTC actual use study in pharmacy sites where the principal investigator will be a pharmacist.

ELIGIBILITY:
INCLUSION CRITERIA

To be eligible for participation, consumers must:

* Male or female, 18 years of age or older
* Select and purchase the study medication for their own use
* Be able to take part in periodic telephone interviews regarding their use of and experience with the medication
* Give written informed consent for participation

EXCLUSION CRITERIA Consumers will be excluded from participation if they meet any of the following criteria:

* Allergic to rabeprazole
* Currently have trouble or pain swallowing food
* Currently have vomiting with blood
* Currently have bloody or black stool
* Currently pregnant or breast-feeding
* Participated in a study regarding a heartburn medication during the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2006-04; Study Completion 2007-01

PRIMARY OUTCOMES:
The percentage of subjects who make an appropriate initial decision about whether to select AcipHex. OTC for their own use | screening visit (Day 0 )
The percentage of subjects who follow key directions for use (1 tablet per day, 14-day course of treatment, and no more than one course of treatment every 4 months) | 14 day treatment period; up to 4 months
The percentage of subjects who make appropriate ongoing decisions about suitability for treatment (including consulting a physician and appropriately modifying or discontinuing use based on label directions) | 14 day treatment period; up to 4 months
The percentage of subjects who experience serious / non-serious adverse events | : 14 day treatment period; up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cyrille, MD, Study Director — Eisai Inc.
Locations (33):
- United States (33):
  - Civic Center Pharmacy, Scottsdale, Arizona
  - Wynn's Pharmacy, Inc., Griffin, Georgia
  - Monfort Drug Company, Inc., Lawrenceville, Georgia
  - Eckerd Drug #234, Marietta, Georgia
  - The Medicine Shoppe, Kansas Ciry, Kansas
  - Stark Pharmacy, Overland Park, Kansas
  - Goodrich Pharmacy, Andover, Minnesota
  - Goodrich Pharmacy, Anoka, Minnesota
  - Goodrich Pharmacy, Blaine, Minnesota
  - Goodrich Pharmacy, Elk River, Minnesota
  - Goodrich Pharmacy, Saint Francis, Minnesota
  - North Oak Pharmacy, Kansas City, Missouri
  - Stevenson Family Pharmacy, Saint Joseph, Missouri
  - Countryside Pharmacy, Savannah, Missouri
  - Family Prescription Center, Bethlehem, Pennsylvania
  - T.B. Bond Pharmacy, Hillsboro, Texas
  - Studewood Pharmacy, Houston, Texas
  - Kashmere Pharmacy, Houston, Texas
  - Longhorn Drug Company, Kilgore, Texas
  - Louis Morgan Drug #1, Longview, Texas
  - The Medicine Shoppe #1511, Spring, Texas
  - West Houston Pharmacy, Tyler, Texas
  - Mountain View Pharmacy, Bountiful, Utah
  - Gibson United Drug, Murray, Utah
  - Apothecary Shoppe, Salt Lake Ciry, Utah
  - Jolley's Corner Pharmacy #1, Salt Lake City, Utah
  - Family Plaza Pharmacy, West Jordan, Utah
  - Montpelier Pharmacy, Inc., Montpelier, Virginia
  - Lafayette Pharmacy, Richmond, Virginia
  - Rxtracare/U & I Pharmacy, Bellevue, Washington
  - Ostrom Drugs, Kenmore, Washington
  - Manhattan Drug, Seattle, Washington
  - Kusler's Pharmacy, Snohomish, Washington